CLINICAL TRIAL: NCT03749512
Title: Preoperative Neutrophil-lymphocyte Count Ratio in Prediction of the Grade of Lung Tumor.
Brief Title: NLCR in Prediction of the Grade of Lung Tumor.
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: NLCR-01
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Lung Neoplasm
Keywords: NLCR, The neutrophil-lymphocyte count ratio, Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Group of patients with lung tumor qualified for thoracic surgery intervention with routine, preoperative complete blood count test and routine postoperative histopathological examination of lung tumor.
  Interventions: Diagnostic Test: Complete blood count; Other: Histopathological examination

INTERVENTIONS:
Diagnostic Test: Complete blood count — During routine preoperative blood test complete blood count is taken.
Other: Histopathological examination — Routine postoperative histopathological examination of lung tumor.

SUMMARY:
The aim of the study is to assess whether the value of neutrophil-lymphocyte count ratio from the routine preoperative blood test may predict lung tumors' grading.

DETAILED DESCRIPTION:
Lung cancer remains as one of the leading causes of death among oncology patients. Close connection between inflammation and pathogenesis of some neoplasms was determined in a number of studies. Some studies show promise that ratio of neutrophil to lymphocyte count (NLCR) may be recognized as a prognostic marker for several carcinomas: renal, lung and colorectal. The aim of the study is to assess whether the value of neutrophil-lymphocyte count ratio from the routine preoperative blood test may predict lung tumors' grading. During routine preoperative blood tests complete blood count is done and NLCR, WBC, neutrophil and lymphocyte count is noted. After the thoracic surgery intervention and histopathological examination grading of lung tumor is noted.

ELIGIBILITY:
Inclusion Criteria:

* consecutive thoracic surgery patients with lung cancer grading confirmed by histopathology postoperatively
* preoperative routine complete blood count analysis

Exclusion Criteria:

* infectious disease
* pregnancy
* autoimmunologic disease
* other known conditions or treatments that may influence the blood count (seropositivity for HIV, chemotherapy, and corticotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive thoracic surgery patients admitted to SPSK nr 1 in Zabrze between October 2014 and October 2018 with lung tumor qualified for thoracic surgery intervention
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Neutrophil-lymphocyte count ratio | From October 1, 2014 to October 15, 2018
  Neutrophil-lymphocyte count ratio is measured during routine preoperative blood tests.

SECONDARY OUTCOMES:
Neutrophil count | From October 1, 2014 to October 15, 2018
  Neutrophil count is measured during routine preoperative blood tests.
Lymphocyte count | From October 1, 2014 to October 15, 2018
  Lymphocyte count is measured during routine preoperative blood tests.
Leucocyte count | From October 1, 2014 to October 15, 2018
  Leucocyte count is measured during routine preoperative blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiołek, MD PhD, Study Chair — Medical University of Silesia
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland